CLINICAL TRIAL: NCT06452433
Title: Gumarontinib Combined With Third-generation EGFR-TKI in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer With MET Amplification Following EGFR-TKI Treatment Failure.
Brief Title: Gumarontinib Combined With 3rd EGFR-TKI in Patients With Non-small Cell Lung Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jie Wang, Chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-HYT-NSCLC-K03
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — glumetinib; osimertinib; aumolertinib; aflutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gumarontinib combined with third-generation EGFR-TKI (Experimental): Patients were treated with Gumarontinib in combination with third-generation EGFR-TKI (Osmertinib,Almonertinib, Furmonertinib) oral therapy until disease progression or the onset of intolerable toxicity, treatment is expected to last 3-6 months.
  Interventions: Drug: gumarontinib; Drug: third-generation EGFR-TKI (Osimertinib, Almonertinib or Furmonertinib)

INTERVENTIONS:
Drug: gumarontinib — 300 mg , qd ,po, expect 6 months.
  Other Names: SCC244
Drug: third-generation EGFR-TKI (Osimertinib, Almonertinib or Furmonertinib) — According to the actual situation of patients. Take as recommended, expect 6 months.
  Other Names: third-generation EGFR-TKI

SUMMARY:
This study evaluated the efficacy and safety of gumarontinib combined with third-generation EGFR-TKI in the treatment of locally advanced or metastatic NSCLC with MET amplification after first-line EGFR-TKI failure, without limiting the type of third-generation EGFR-TKI. The study was divided into 2 cohorts: Cohort 1 included patients with MET amplification after third-generation EGFR-TKI first-line therapy resistance, and cohort 2 included patients with MET amplification after first-generation EGFR-TKI first-line therapy resistance.

DETAILED DESCRIPTION:
This study evaluated the efficacy and safety of gumarontinib combined with third-generation EGFR-TKI in the treatment of locally advanced or metastatic NSCLC with MET amplification after first-line EGFR-TKI failure, without limiting the type of third-generation EGFR-TKI. The study was divided into 2 cohorts: Cohort 1 included patients with MET amplification after third-generation EGFR-TKI first-line therapy resistance, and cohort 2 included patients with MET amplification after first-generation EGFR-TKI first-line therapy resistance. Patients will receive the combination until disease progression or intolerable toxicity. A total of 91 patients who met the inclusion and exclusion criteria were included in the study. The primary endpoint was ORR.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* Locally advanced or metastatic (stage IIIB-IV) NSCLC confirmed histologically or cytologically, stage III patients are unresectable and are not suitable for radical concurrent chemoradiotherapy.
* ECOG 0~1.
* Expected survival time ≥3 months
* Patients with EGFR mutations known to be associated with drug sensitivity (i.e., exon 19 deletion or L858R mutation).
* For advanced NSCLC, 2 or 3 generations of EGFR-TKI or EGFR-TKI (EGFR-TKI monotherapy, combination chemotherapy or bevacizumab are acceptable) have been treated with treatment failure, and EGFR-TKI has only been received as first-line therapy: Cohort 1: Third-generation EGFR-TKI therapy failed (EGFR-TKI monotherapy, combination chemotherapy, or bevacizumab could be used) without first - or second-generation EGFR-TKI therapy; Cohort 2: EGFR-TKI therapy failed in the first or second generation (EGFR-TKI monotherapy, combination chemotherapy, or bevacizumab were acceptable), and the status of T790M was not limited without the third generation of EGFR-TKI therapy or the first three generations of EGFR-TKI therapy < 4 weeks (28 days);
* Met the following criteria for EGFR-TKI treatment failure (acquired resistance): Continuous treatment with EGFR-TKI in the past; Treatment with EGFR-TKI resulted in any of the following objective clinical benefits (RECIST 1.1) ; Documented partial or complete remission; Clinical benefit for ≥6 months; Imaging disease progression during EGFR-TKI treatment (RECIST 1.1).
* Specimens collected after treatment with EGFR-TKI for disease progression meet criteria for MET amplification (FISH GCN≥5 or MET/CEP7≥2, or NGS GCN≥2.3).
* At least one measurable lesion according to RECIST 1.1 criteria.
* Has recovered from adverse effects of any prior chemotherapy, surgery, radiation, or other antitumor therapy to CTCAE 5.0 ≤ Grade 1 or baseline (except for toxicities such as hair loss that the investigator determines are not a safety risk).
* Normal bone marrow and organ function: Neutrophils (ANC) ≥1.5×10^9/L, platelets (PLT) ≥90×10^9/L, hemoglobin (Hb) ≥90g/L,patients whose hematological indexes were at a critical value and could not meet the above criteria were determined by the investigator according to the patient's physical condition; AST, ALT and alkaline phosphatase (ALP) were all ≤2.5× upper limit of normal range (ULN), and ≤5×ULN when liver metastases occurred;Total bilirubin ≤1 x ULN or ULN < total bilirubin ≤1.5 x ULN, and AST≤1 x ULN; Creatinine clearance >50 ml/min (calculated according to Cockroft-Gault)
* Patients were fully aware of and volunteered to participate in the study.

Exclusion Criteria:

* Patients who had previously been treated with MET inhibitors.
* In addition to EGFR and MET, have gene mutations sensitive to other targeted drugs such as ALK and ROS1.
* Patients who have previously received EGFR-TKI rechallenge therapy.
* Study patients with neurologically unstable CNS metastases in the central nervous system who had symptoms related to brain metastases prior to treatment initiation, or who required increased steroid doses to control CNS disease (patients with controlled CNS metastases may participate in this trial).
* The following medications are required 2 weeks prior to and during study therapy: drugs that may lead to prolonged QTc interval or tip torsive ventricular tachycardia, transporter MATE1, MATE2K substrate, and strong inducers of CYP3A4.
* Present or past 5 years with other malignancies (except cured skin basal cell carcinoma, carcinoma in situ, etc.).
* Received other antitumor agents (except EGFR-TKI) within 5 half-lives prior to initial administration of the investigational drug; If the patient's last anti-tumor treatment prior to screening was third-generation EGFR-TKI, the patient may continue to receive third-generation EGFR-TKI until admission to the regimen without medication interruption.
* Adverse effects did not recover after receiving extensive radiation therapy within 4 weeks of study treatment initiation or palliative local radiation therapy within 1 week of study treatment initiation.
* Interstitial lung disease (ILD) or pneumonia requiring systemic steroid treatment.
* Study received major surgery or significant trauma within 4 weeks before the start of treatment.
* Hyperkinetic/venous thrombotic events or embolic events, such as stroke (including transient ischemic attack), deep vein thrombosis, pulmonary embolism, occurred within 6 months before the first dose;
* Patients with dysphagia, complete or incomplete digestive obstruction, active gastrointestinal bleeding, perforation, etc. affecting oral drug absorption (frequent vomiting, diarrhea, etc.);
* In the 6 months prior to screening, cardiovascular disease met any of the following criteria: a) congestive heart failure ≥3 of the New York College of Cardiology (NYHA); Or left ventricular ejection fraction (LVEF) < 50%; b) severe arrhythmias requiring medical treatment; c) Screening period mean resting corrected QT interval (QTcF) > 470 ms for women or >450 ms for men (using the Fridericia formula [QTc = QT/(RR^0.33)], averaging results from three 12-lead ECG tests), or the presence of a risk factor for tip torsion ventricular tachycardia, For example, a family history of hypokalemia, long QT syndrome, or familial arrhythmia judged by the investigator to be clinically significant; d) Uncontrolled hypertension (defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg after treatment with standardized antihypertensive drugs); e) acute myocardial infarction, severe or unstable angina pectoris, coronary or peripheral artery bypass grafting within 6 months prior to initial administration; f) Clinically significant arrhythmias.
* An active, uncontrolled bacterial, viral, or fungal infection requiring systemic treatment, defined as persistent signs/symptoms associated with the infection that do not improve despite the use of appropriate antibiotics, antiviral therapy, and/or other treatment;
* Patients with active hepatitis B (HbsAg or HBcAb positive and HBV DNA higher than the upper limit of normal), active hepatitis C (HCV antibody positive and HCV RNA higher than the upper limit of the study center), HIV antibody positive;
* Known allergy or intolerance to therapeutic drugs or their excipients;
* Pregnant or lactating women;
* The investigator believes that the subjects are not suitable to participate in this clinical study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2027-12-12 (Estimated); Study Completion 2028-02-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From initial medication to the date of first documented progression or end of medication. Assessed up to 6 months.
  To investigate antitumor efficacy of study, proportion of patients with complete (CR) or partial response (PR).

SECONDARY OUTCOMES:
Disease control rate | From initial medication to the date of first documented progression or end of medication, whichever came first, assessed up to 6 months.
  To investigate antitumor efficacy of study, proportion of patients with complete , partial or stable response (SD).
Duration of response | from first achieving CR or PR to the onset of disease progression (PD) or death, whichever occurs first, Assessed up to 36 months.
  Time from first achieving CR or PR to the onset of disease progression (PD) or death, whichever occurs first
Progression free survival | From initial medication to the date of first documented progression or end of medication, whichever came first. Assessed up to 24 months.
  To investigate antitumor efficacy of study. From initial medication to the date of first documented progression or end of medication, whichever came first.
Overall survival | From initial medication to the date of death from any cause. Assessed up to 36 months.
  To investigate antitumor efficacy of study. From initial medication to the date of death from any cause.
Incidence of adverse events and severity of adverse events as assessed by CTCAE 5.0 | Assessed except to 10 months.
  To assess the incidence and severity of adverse events in combination regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences